CLINICAL TRIAL: NCT00873470
Title: Long Term Evolution of the Anterograde Refractory Period of Accessory Duct in the Wolff-Parkinson-White Syndrome
Brief Title: Wolff-Parkinson-White Syndrome Anterograde Refractory Period of Accessory Duct
Acronym: WPW
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BRD 08/9-I
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Wolff-Parkinson-White Syndrome
MeSH Terms: conditions — Wolff-Parkinson-White Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stimulation (Experimental): All patients included have the stimulation
  Interventions: Procedure: esophagal stimulation

INTERVENTIONS:
Procedure: esophagal stimulation — ECG (rest) esophagal stimulation (rest and during effort)

SUMMARY:
The study consists of the realization of a new esophageal stimulation for patients already stimulated 10 years ago.

The investigators would like to make a long term evaluation of the evolution of anterograde effective refractory period of accessory duct in the WPW syndrome.

This study will be realized by esophageal stimulation.

ELIGIBILITY:
Inclusion Criteria:

* 21 < age < 64 years
* First esophagal stimulation with evaluation of effective anterograde refractory period > 10 years
* Informed consent signed
* Diagnosis of Wolff-Parkinson-White syndrome
* No procedure of ablation of accessory duct

Exclusion Criteria:

* Ablation of accessory duct
* Patient with contraindication to esophageal stimulation
* Patient with contraindication to effort test

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measurement of effective anterograde refractory period of accessory duct and its evolution for a follow up superior to 10 years | Day 0

SECONDARY OUTCOMES:
Triggering a supra-ventricular tachycardia during the stimulation. | Day 0
Presence of symptoms linked to WPW syndrome during the interval separating the 2 esophageal stimulation. | Day 0

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes UH, Nantes, France